CLINICAL TRIAL: NCT00910442
Title: The Effect of Substrate Supply on Modulating Plasma GSH Levels in Treated HIV+ Patients
Brief Title: Glutathione and Its Precursors in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Roberto Carlos Burini, UNESP Faculdade de Medicina de Botucatu
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-24
Record Dates: First submitted 2009-05-27; First posted 2009-05-29 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Glutamine; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Group (Experimental): Dietary supplement:N-acetylcysteine 1g/day and Glutamine 20g/day for 7 consecutive days. The dietary supplements were intermediated by 7 days of washout with usual diet.
  Interventions: Dietary Supplement: Glutathione precursors
- Control Group (Active Comparator): Healthy HIV negative subjects submitted to the same dietary supplement than experimental group: N-acetylcysteine 1g/day and Glutamine 20g/day for 7 consecutive days. The dietary supplements were intermediated by 7 days of washout with usual diet.
  Interventions: Dietary Supplement: Glutathione precursors

INTERVENTIONS:
Dietary Supplement: Glutathione precursors — HIV+ patients were assigned to 7 day diets containing either NAC or Gln
  Other Names: Glutamine (L-glutamine); NAC (N-acetyl-L-cysteine)

SUMMARY:
The aim of this study is to investigate the responses of the serum amyloid A (SAA) pathway to dietary supplements of glutamine (Gln) and cysteine (Cys) together with methionine (Met)-overloading in HIV+ patients comparatively to healthy controls.

DETAILED DESCRIPTION:
Introduction: Among the 4 sulphur-containing amino acids (SAA), only Met and Cys are incorporated into proteins, but Hcy and Tau are related to oxidative stress and glutathione (GSH), the major intracellular hydro-soluble anti-oxidant agent. HIV+ patients present low levels of antioxidant nutrients, including GSH and its precursors.

Objective: To investigate the responses of the SAA pathway to dietary supplements of Gln and Cys together with Met-overloading in HIV+ patients comparatively to healthy controls.

Methods: Twelve HIV+ (6 males and 6 females, 25-36 yrs old) patients under HAART (one HIV protease inhibitor in combination with two nucleoside analogs) for at least one year and 20 (10M and 10F, 23-28 yrs old) healthy controls were randomly assigned to 7-day diets containing either NAC (N-acetylcysteine, 1g/d) or Gln (20g/d), with a 7-day washout period with their usual diet (UD). Blood samples were drawn after overnight fast before and after (2h and 4h) ingesting the Met (100 mg/kg) overload (Met-OL) with determination of the area under the curve (AUC). HPLC plasma analysis of SAA (Met, Hcy, Cys and Tau), GSH and GSSG and Ser, Gly, Glu and Gln was carried out at moments before (MO) and after 7-day diets (M1). Additionally, at baseline, both groups were assessed for anthropometry (BMI, kg/m2; body fat %) and plasma biochemistry (creatinine, urea, γ-glutamyl transpeptidase, glucose, triglycerides, cholesterol, uric acid, albumin, folic acid and vitamin B12).The HIV+ group (G2) was also characterized by the viral load, CD4+ and CD8+ lymphocytes counts. Statistical comparisons were undertaken among diets between groups with p = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* antiretroviral therapy for at least one year

Exclusion Criteria:

* presence of any renal or liver failure
* ingestion of either vitamins B or GSH precursors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-02; Primary Completion 2007-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Plasma glutathione | 7 days

SECONDARY OUTCOMES:
Plasma sulfur amino acids | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Roberto C Burini, PhD, Principal Investigator — UNESP Medical School

REFERENCES:
- [Derived] Burini RC, Borges-Santos MD, Moreto F, Yu YM. Comparative effects of acute-methionine loading on the plasma sulfur-amino acids in NAC-supplemented HIV+ patients and healthy controls. Amino Acids. 2018 May;50(5):569-576. doi: 10.1007/s00726-018-2538-2. Epub 2018 Feb 1. PMID 29392418
- [Derived] Borges-Santos MD, Moreto F, Pereira PC, Ming-Yu Y, Burini RC. Plasma glutathione of HIV(+) patients responded positively and differently to dietary supplementation with cysteine or glutamine. Nutrition. 2012 Jul;28(7-8):753-6. doi: 10.1016/j.nut.2011.10.014. Epub 2012 Jan 20. PMID 22261571